CLINICAL TRIAL: NCT06886165
Title: My Avenue to helP - Adaptive Mentalization-based Integrative Treatment Compared to Management as Usual for Youths With Multiple Problems: a Non-Randomized Controlled Feasibility Trial
Acronym: MAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pia Jeppesen (Other)
Collaborators: Lejre Municipality (Unknown); Roskilde Municipality (Unknown); Child and Adolescent Mental Health Services, Region Zealand (Unknown); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor-Investigator, Pia Jeppesen, Professor, PhD, Head of Research, Department of Child and Adolescent Psychiatry, Psychiatric Research Unit, Region Zealand, Denmark
Organization: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-1084; P-2024-17167 (Other: Region Zealand)
Record Dates: First submitted 2025-02-21; First posted 2025-03-20 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Care; AMBIT; Adaptive Mentalization-Based Integrative Treatment; Child and Adolescent Psychiatry; Health Care Professionals; Mental Health Services; Community Mental Health Services; Emergency Services, Psychiatric; Social Work, Psychiatric
Keywords: AMBIT; Adative Mentalization-Based Integrative Treatment; Child and Adolescent Psychiatry; Cross-sectoral Collaboration; Interdisiplinary Collaboration; Implementation; Municipalities; Mentalization; Social Functioning; CAMHS; Feasibility Study; Primary Health Care; Child and Adolescent Mental Health Services
MeSH Terms: conditions — Social Adjustment | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MAP intervention (Experimental): Participants in the experimental arm of the MAP-Project will receive one year of treatment with the MAP-intervention.
  Interventions: Behavioral: My Avenue to HelP
- Management as Usual, MAU (Active Comparator): Management as Usual will be carried out in the diverse municipalities of residence of the control and the Child and Adolescent Mental Health Services in Region Zealand.
  Interventions: Behavioral: Management as Usual

INTERVENTIONS:
Behavioral: My Avenue to HelP — The MAP intervention is based on AMBIT principles. A MAP team, consisting of designated employees from CAMHS and two municipalities, will be trained in AMBIT. A Key-Worker and a Mentalizing Case Manager will be assigned to each participant and step into the existing network, taking responsibility for integrating AMBIT principles into all aspects of the work with and around the young person. The Key-worker from the MAP team is responsible for reaching out to the young person at least once a week during the intervention. The Mentalizing Case Manager ensures that mentalization is upheld in the professional network. CAMHS will offer treatment as usual in accordance with the existing evidence-based clinical guidelines and best practice for any specific mental health disorder.
  The MAP team members will meet once a week to work as a team and collaborate closely with family members and other potential informal caregivers. The network of helpers will meet and coordinate monthly.
  Arms: MAP intervention
Behavioral: Management as Usual — Participants in the control group will receive non-manualized, standard treatment in CAMHS in collaboration with their municipality of residence, following local practice and guidelines. The MAU will be slightly enhanced compared to standard treatment: a) the young people will have an open case file during one year of participation in the MAP project (and longer if indicated), and b) the standard care services will receive feedback from the research assessment at baseline (after approval of the specific content from parents and the young person) in order to help the young person's caseworker to coordinate the support. These enhancements are made to improve the cohesion of care for the young person, yet without applying the mentalization-based AMBIT principles and MAP teams of the MAP treatment condition.
  principles applied in the MAP treatment condition.
  Arms: Management as Usual, MAU

SUMMARY:
My Avenue to HelP (MAP) is a non-randomized feasibility study testing the implementation of a cross-sectoral collaboration targeted youths, aged 12-17 years, with multiple social and psychological problems. MAP is a one-year intervention based on Adaptive Mentalization-Based Integrative Treatment (AMBIT). MAP is not a new treatment method, but rather a new way of offering and organizing support in the existing network around the young person. The objective is to create a new way for professionals across sectors to collaborate in supporting our most vulnerable youth. Thereby, the investigators aim to benefit the youths by incorporating a mentalizing stance to promote lasting changes beyond the intervention period. The MAP Project will run from 2025 to 2027.

The research will consist of two work packages (WPs)

* WP1 will test the feasibility of the MAP project examining a) whether young people can be successfully recruited to the project b) if the evaluation design and methods are feasible and c) if the intervention is feasible to participants and employees (quantitatively).
* WP2 will assess implementation determinants and evaluate the implementation strategies employed in the project. Furthermore, the acceptability of the intervention will qualitatively be assessed by interviews with selected participants, their parents, as well as employees.

Participants:

In total 60 youths aged 12-17 years from Region Zealand, Denmark:

* 40 youths will be enrolled and receive the one-year MAP Intervention; 30 youths residing in Roskilde Municipality and 10 residing in Lejre Municipality
* 20 youths from other municipalities in Region Zealand will be included in the trial as a control group.

To assess the nature and extent of the mental health problems and potential psychiatric disorders among the participating youths, the parents and the young person will be asked to complete an online questionnaire (Development and Well-Being Assessment (DAWBA)).

ELIGIBILITY:
Inclusion Criteria:

* Criterium A) Documented record of multiple problems defined as at least 2 of the following: (i) Absence from school / non-adherence to education (ii) Risk behaviors like alcohol or cannabis abuse, or repeated suicide attempts or self-harm requiring somatic treatment.(iii) Repeated visits at emergency-, trauma-, or acute wards. And/or one of the following: (iv) Contact with police or legal justice system. (v) Homelessness within the last year.
* Criterium B) Age 12-17 years at time of inclusion.
* Criterium C) Strong indication of mental disorders defined as a diagnosis of a mental disorder. The type of mental disorders will be further substantiated using the DAWBA after recruitment (Goodman et al., 2000).
* Criterium D) Written/signed informed consent from all legal guardians (in most cases both parents) and oral consent from youths aged 15 years and older. Written/signed informed consent from the youths themselves will be collected when they turn 18 if they do so during the study period.

Exclusion Criteria:

* Indications of substantial intellectual disability corresponding to IQ below 50, or a level of daily and social functions that do not enable participation in research (e.g., if the young person is not deemed to have the capacity to understand the implications of the study and provide oral consent).
* Not living in Region Zealand.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcome 1: Recruitment | 8 weeks after the last patient is enrolled
  Feasibility outcome 1 will be assessed by calculating the proportion of families that accept inclusion out of those who fulfill inclusion criteria. The intervention will be deemed acceptable if ≥50% of the families that are eligible (assessed at an informational meeting) also consent to participate in the MAP study.
Feasibility Outcome 2: Adherence to treatment protocol | Weekly registration of the contact between the young person and the keyworker from baseline and during the complete 52 weeks of intervention.
  Feasibility outcome 2 will be assessed by contacting the Keyworker monthly to inquire about the contacts made/attempted by the Keyworker to the young person/network around the young person. Type of contact made between the Keyworker and the young person, and alternatively whom the Keyworker was in contact with within the indigenous network of the young person, in cases where the young person does not want direct contact with the Keyworker, will be registered as well. The intervention will be deemed acceptable if ≥70% of youths in the MAP intervention do not experience a pause of 4 continuous weeks between contacts.
Feasibility Outcome 3: Satisfaction with the intervention | Assessment within + / - 2 weeks after end of treatment
  Feasibility outcome 3 regarding the satisfaction with treatment in MAP will be assessed using item 16.4 of the Client Satisfaction Questionnaire. The intervention will be deemed acceptable if ≥70% of youths and parents would recommend MAP to a friend.
Feasibility Outcome 4: Satisfaction with the intervention | Assessment within 2 weeks after the intervention period ends.
  Feasibility outcome 4 will be assessed by a questionnaire developed for the MAP project and will be delivered to all workers (in the MAP teams) and leaders involved in MAP in Roskilde, Lejre, and CAMHS. The intervention will be deemed acceptable if >70% of MAP team staff and leaders will continue to prioritize the intervention.
Feasibility Outcome 5: Reliability of the measurement of change in youth's social function | Assessment within 2 weeks after the intervention period ends.
  Feasibility outcome 5 will be deemed acceptable if ≥70% of youths who consented to participate in the MAP project, participated in the 'Personal and Social Performance Scale Interviews at baseline and after 1 year.

OTHER OUTCOMES:
Primary exploratory outcome: Change in youths' social function | The PSP interview will be conducted at baseline and at end of intervention (after 52 weeks, +/- 14 days).
  Change in youths' social function covering four domains (socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors, measured with the Personal and Social Performance (PSP) Scale, rated by researchers using multiple sources of information. Overall functioning will be scored on a scale from 0 (minimum value [worst outcome], complete lack of autonomy) to 100 (maximum value [best outcome], excellent functioning).
Monitoring of adverse events | Weekly screening for adverse events during the complete 52 weeks treatment.
  We anticipate no or minimal adverse effects or adverse events related to the AMBIT and MAU interventions in the trial. The independent observer will be responsible for the recording and classification of events based on the weekly contact with the participants and surveillance of the electronic health record system (Sundhedsplatformen) to cover adverse events according to the following definitions:
  Adverse Event (AE): any undesirable medical event occurring to a participant during a clinical trial, which does not necessarily have a causal relationship with the intervention.
  Adverse Reaction (AR): any undesirable and unintended medical response related to the intervention occurring to a participant during a clinical trial.
  Serious Adverse Event (SAE): any adverse event that results in death, is life-threatening, requires hospitalization or prolongation of existing hospital stay
Secondary exploratory outcomes: Participation in education, employment, or training in the past four weeks | The assessment will be conducted at baseline and at end of treatment (after 1 year, +/- 14 days).
  Participation in education, employment, or training in the past four weeks, rated by an independent observer based on multiple sources of information from a short interview in connection with the Personal and Social Performance Scale assessment.
Secondary exploratory outcomes: Change in well-being | The questionnaire is administered to the young person and the primary parent/caregiver at baseline, midway (after 182 days +/- 14 days), and after 1 year (365 days +/- 30 days) to measure changes before, during, and after the treatment period.
  Change in well-being, self-reported with the WHO-5 well-being index. The WHO-5 includes 5 questions scored on a Likert scale from 0 (low well-being) to 5 (high well-being) resulting in a sum score of 0 to 25.
Secondary exploratory outcomes: Change in personal recovery | The questionnaire is administered to the young person and the primary parent/caregiver at baseline, midway (after 182 days +/- 14 days), and after 1 year (365 days +/- 30 days) to measure changes before, during, and after the treatment period.
  Change in personal recovery, self-reported, measured by the Brief INSPIRE-O, which has recently been validated in a Danish context. The Brief INSPIRE-O includes 5 questions scored on a Likert scale from 0 (low well-being) to 4 (high well-being) resulting in a sum score of 0 to 20.
Secondary exploratory outcomes: Change in health-related quality of life | The questionnaire is administered to the young person and the primary parent/caregiver at baseline, midway (after 182 days +/- 14 days), and after 1 year (365 days +/- 30 days) to measure changes before, during, and after the treatment period.
  Change in health-related quality of life measured by the Child Health Utility 9D (CHU9D), self- and parent-reported. All nine items of the CHU9D have five unnumbered response options which are converted to scores of 1-5, resulting in a sum score of 9 to 45. The instrument allows for the calculation of Quality-Adjusted Life Years (QALYs). It is a measure used to assess how many good life years are gained or lost by introducing new health technology or organization.
Secondary exploratory outcomes: Mental health problems and disorders | The questionnaire is administered to the young person and the primary parent/caregiver at baseline, midway (after 182 days +/- 14 days), and after 1 year (365 days +/- 30 days) to measure changes before, during, and after the treatment period.
  Mental health problems and disorders measured by the Strengths and Difficulties Questionnaire (SDQ) (Goodman, 1999), self- and parent-reported. The SDQ contains 25 items, which cover five subscales relating to the children's emotional problems, peer problems, behavioral problems, hyperactivity and pro-social behavior. Responses to the subscales on emotional problems, peer problems, behavioral problems, and hyperactivity can be used to calculate a total difficulties score. Each subscale score ranges from 0-10, implying that the total difficulties score ranges from 0 to 40 An impact score is calculated from five items; whether the difficulties upset or distress the child and how much the difficulties interfere with home life, friendships, classroom learning, and leisure activities. Each item is scored on a scale from 0 to 10. To score 1 or 2, the interference from the difficulties in that domain must be assessed to either "quite a lot" or "a great deal", resulting in an impact score.
Secondary exploratory outcomes: Participant satisfaction | The questionnaire is administered to the participant at the end of intervention (after 52 weeks + / - 2 weeks)
  Participant satisfaction measured with the Client Satisfaction Questionnaire, self-reported. The scale consists of 8 questions scored on a 4-point Likert Scale ranging from low to high satisfaction with different aspects of the intervention. The total score ranges from 8 (minimum value [bad outcome], low satisfaction) to 32 (maximum value [good outcome], high satisfaction).
Secondary exploratory outcomes: Parental satisfaction | The questionnaire is administered to the primary parent/caregiver at the end of intervention (after 52 weeks + / - 2 weeks)
  Parental satisfaction and experience with the treatment of their child will be measured with the Experience of Service Questionnaire. The scale consists of 10 questions scored on a 3-point Likert Scale. The total score ranges from 0 (minimum value [bad outcome], poor satisfaction]) to 20 (maximum value [good outcome], high satisfaction]).
Secondary exploratory outcomes: Adherence to planned care in CAMHS | All planned and completed appointments with CAMHS will be documented by the investigators during the complete 52 weeks of intervention. The investigators will screen for emergency healthcare service use weekly during the complete 52 weeks of intervention
  Adherence to planned care in CAMHS and the use of emergency healthcare will be assessed through information from the young person's patient records.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jeppesen, Professor, MD, Principal Investigator — University of Copenhagen and head of the Research Department in the Child and Adolescent Mental Health Services, Region Zealand; Martin Køster Rimvall, PhD, MD, Principal Investigator — Research Department in the Child and Adolescent Mental Health Services, Region Zealand
Locations (1):
- Child and Adolescent Psychiatric Department, Psychiatry Region Zealand, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The pseudonymous quantitative data can be made available from six months after the publication date of the scientific articles written by the PhD student (from 2029). Proposals for use of data and requests for access should be directed to the principal investigator Pia Jeppesen, mail: pijep@regionsjaelland.dk.
  To gain access, researchers will need to sign a data access agreement with the Department of Child and Adolescent Psychiatry, Copenhagen University Hospital - Psychiatry Region Zealand, Roskilde, Denmark. The pseudonymous individual participant data can be made available to investigators for research that have been approved by independent review committees. The data access will be granted on a case-by-case basis by the principal investigator. Access will be granted to the extent permissible by the General Data Protection Regulation and the Danish Data Protection Act. Making the data available may require approval from the Danish Data Protection Authority.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD including the SAP will become available 6 months after the publication of the summary of all results of the feasibility trial (expected access in 2029). The study protocol will be published during the period of recruitment of participants in 2025-26.
Access Criteria: The IPD and supporting information will be available for researchers upon request for research that have been approved by independent review committees and to the extent permissible by the General Data Protection Regulation and the Danish Data Protection Act. Making the data available may require approval from the Danish Data Protection Authority.
  The pseudonymous quantitative data will be shared electronically in excel sheets.